CLINICAL TRIAL: NCT06625671
Title: A Randomized, Double-Blind, Phase 1/2a Study to Evaluate the Safety, Tolerability, PK and PD of DB-2304 for Injection in Healthy Adult Participants and Participants With Systemic Lupus Erythematosus or Cutaneous Lupus Erythematosus
Brief Title: A Phase 1/2a Study of DB-2304 in Healthy Adults and SLE Participants
Status: Recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: DualityBio Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: Double | Purpose: Treatment
Other Study IDs: DB-2304-101
Record Dates: First submitted 2024-09-20; First posted 2024-10-03 (Actual); Last update posted 2025-12-18 (Actual); Status verified 2025-12

CONDITIONS: Systemic Lupus Erythematosus (SLE)
MeSH Terms: conditions — Lupus Erythematosus, Systemic | interventions — Prednisone

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (8):
- Dose Level 1 (Experimental)
  Interventions: Drug: DB-2304; Drug: Placebo; Drug: Prednisone
- Dose Level 2 (Experimental)
  Interventions: Drug: DB-2304; Drug: Placebo; Drug: Prednisone
- Dose Level 3 (Experimental)
  Interventions: Drug: DB-2304; Drug: Placebo; Drug: Prednisone
- Dose Level 4 (Experimental)
  Interventions: Drug: DB-2304; Drug: Placebo; Drug: Prednisone
- Dose Level 5 (Experimental)
  Interventions: Drug: DB-2304; Drug: Placebo; Drug: Prednisone
- Dose Level 6 (Experimental)
  Interventions: Drug: DB-2304; Drug: Placebo
- Dose Level 7 (Experimental)
  Interventions: Drug: DB-2304; Drug: Placebo
- Dose Level 8 (Experimental)
  Interventions: Drug: DB-2304; Drug: Placebo

INTERVENTIONS:
Drug: DB-2304 — DB-2304
Drug: Placebo — Placebo
Drug: Prednisone — Prednisone
  Arms: Dose Level 1; Dose Level 2; Dose Level 3; Dose Level 4; Dose Level 5

SUMMARY:
A Phase 1/2a Study of DB-2304 in Healthy Participants and Participants with Systemic Lupus Erythematosus or Cutaneous Lupus Erythematosus

ELIGIBILITY:
Inclusion Criteria (Part A):

1. Participants who fully understand the purpose, nature, method, and potential adverse reactions of the study and voluntarily sign the informed consent form (ICF) and agree to participate.
2. Healthy male or female participants; 18 to 55 years of age (both inclusive) on the day of signing ICF; meet the body mass index (BMI) criteria.
3. Based on the investigator assessment, there are no abnormal findings or findings with clinical significance from the medical history consultation, physical examination, vital signs assessment, clinical laboratory tests, and 12-lead ECG.
4. Female participants of childbearing potential or male participants agree to use highly effective contraception during the study.
5. Participants who are willing and able to comply with the prescribed protocol treatment and evaluations

Inclusion Criteria (Part B):

1. Participants who fully understand the purpose, nature, method, and potential adverse reactions of the study and voluntarily sign the informed consent form (ICF) and agree to participate.
2. Participants who are willing and able to comply with the prescribed protocol treatment and evaluations.
3. Male or female participants, 18 to 70 years of age (both inclusive) on the day of signing ICF.
4. Currently receiving a stable SLE/CLE treatment regimen of any medication for a period of at least 1 month prior to randomization.

For SLE： 4. Meet the European Alliance of Associations for Rheumatology (EULAR)/American College of Rheumatology (ACR) 2019 classification criteria for SLE.

5. History or presence at Screening of positive antinuclear antibodies (ANA) or anti-double-stranded DNA (anti-dsDNA) antibodies.

6. At screening have active lupus skin disease defined by the SELENA-SLEDAI at screening and randomization.

For CLE： 8. Must have diagnosis of CLE that has been histologically confirmed, with or without systemic LE manifestations.

9.Must have active CLE despite an adequate trial of conventional therapies.

Exclusion Criteria (Part A):

1. Evidence or history of clinically significant diseases.
2. History of herpes zoster (shingles) or recurrent herpes simplex (e.g., oral cold sores or gen-ital sores).
3. Any active or suspected bacterial, viral, fungal, or parasitic infection within 30 days prior to dosing.
4. History of sensitivity to any ingredients of DB-2304.
5. Participants who have undergone surgery within the past 3 months or have plans for sur-gery during the study.

Exclusion Criteria (Part B):

1. Have active lupus nephritis or moderate-to-severe or chronic kidney disease
2. Have active neuropsychiatric SLE within 8 weeks prior to screening
3. Any active skin conditions or active arthritis other than SLE that may interfere with skin or arthritis assessments (e.g., psoriasis, non-LE skin lesions, non-LE alopecia areata, drug-induced lupus, rheumatoid arthritis) at screening.
4. History of, or ongoing, malignant disease, including solid tumors and hematologic malignancies with the exception of basal cell carcinomas and squamous cell carcinomas and carcinoma in situ of the cervix that have been completely excised and considered cured >2 years prior to Screening.
5. Known history of a primary immunodeficiency (e.g., common variable immunodeficiency syndrome), splenectomy, or any underlying condition that predisposes the participant to infection.

NOTE: Other protocol defined Inclusion/Exclusion criteria may apply.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 148 (Estimated)
Dates: Start 2024-10-04 (Actual); Primary Completion 2026-03-23 (Estimated); Study Completion 2026-06-05 (Estimated)

PRIMARY OUTCOMES:
TEAEs | Up to 112 days after last study treatment administration for Part A, and up to 196 days after last study treatment administration for Part B
  Treatment-emergent adverse events
SAEs | Up to 112 days after last study treatment administration for Part A, and up to 196 days after last study treatment administration for Part B
  serious adverse events
ECG parameters | Up to 112 days after last study treatment administration for Part A, and up to 196 days after last study treatment administration for Part B
  12-lead electrocardiograms parameters including HR, PR, QT intervals, QTcF intervals for Fredericia's formula-QT corrected interval), and QRS duration should be determined.
Weight measurements | Up to 112 days after last study treatment administration for Part A, and up to 196 days after last study treatment administration for Part B
  Change and Rate of Change from Baseline in weight
Heart Rate measurements | Up to 112 days after last study treatment administration for Part A, and up to 196 days after last study treatment administration for Part B
  Change and Rate of Change from Baseline in heart rate
Pulse rate measurements | Up to 112 days after last study treatment administration for Part A, and up to 196 days after last study treatment administration for Part B
  Change and Rate of Change from Baseline in pulse rate
Respiratory rate measurements | Up to 112 days after last study treatment administration for Part A, and up to 196 days after last study treatment administration for Part B
  Change and Rate of Change from Baseline in respiratory rate
Body temperature measurements | Up to 112 days after last study treatment administration for Part A, and up to 196 days after last study treatment administration for Part B
  Change and Rate of Change from Baseline in body temperature

CONTACTS AND LOCATIONS:
Overall Officials: Lily Hu, Study Director — DualityBio Inc.
Locations (4):
- United States (3):
  - US03-0, Clearwater, Florida
  - US04-0, Irving, Texas
  - US02-0, San Antonio, Texas
- Site AUS01-0, Melbourne, Victoria, Australia

IPD SHARING:
Plan to Share IPD: Undecided